CLINICAL TRIAL: NCT04558268
Title: Low Dose Prednisone Therapy in Women With Recurrent Pregnancy Loss
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Soroka University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SOR-0461-18-CTIL
Record Dates: First submitted 2020-05-12; First posted 2020-09-22 (Actual); Last update posted 2020-09-22 (Actual); Status verified 2020-02

CONDITIONS: Recurrent Pregnancy Loss(RPL); Recurrent Miscarriage
Keywords: Recurrent pregnancy loss(RPL); Recurrent miscarriage; Prednisone; Autoimmune antibodies; Life birth rate
MeSH Terms: conditions — Abortion, Habitual | interventions — Prednisone; Progesterone; Iron-Dextran Complex; Folic Acid

STUDY DESIGN:
Intervention Model Description: two groups. a treatment group and a placebo group
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- treatment group (Experimental)
  Interventions: Drug: Prednisone; Drug: Progesterone; Dietary Supplement: vit D; Dietary Supplement: Iron Supplement; Dietary Supplement: Folic Acid
- placebo group (Placebo Comparator)
  Interventions: Drug: Progesterone; Dietary Supplement: vit D; Dietary Supplement: Iron Supplement; Dietary Supplement: Folic Acid

INTERVENTIONS:
Drug: Prednisone — Prednisone is a corticosteroid. It prevents the release of substances in the body that cause inflammation. It also suppresses the immune system.
  Prednisone is used as an anti-inflammatory or an immunosuppressant medication. Prednisone treats many different conditions such as allergic disorders, skin conditions, ulcerative colitis, arthritis, lupus, psoriasis, or breathing disorders.
  Arms: treatment group
Drug: Progesterone — Progesterone is a female hormone important for the regulation of ovulation and menstruation.
  Progesterone is used to cause menstrual periods in women who have not yet reached menopause but are not having periods due to a lack of progesterone in the body. It is also used to prevent overgrowth in the lining of the uterus in postmenopausal women who are receiving estrogen hormone replacement therapy.
Dietary Supplement: vit D — Vitamin D acts on our bones, intestines, kidneys and parathyroid glands to keep calcium in balance throughout our body. Vitamin D receptors are also located within our cardiovascular system, lungs, pancreas, skeletal muscle, skin, and reproductive organs. In summary, vitamin D is a prohormone that is essential for good health.
Dietary Supplement: Iron Supplement — Iron is one of the minerals in the human body. It is one of the components of hemoglobin, the substance in red blood cells that helps blood carry oxygen throughout the body.
Dietary Supplement: Folic Acid — Folic acid is a type of B vitamin that is normally found in foods such as dried beans, peas, lentils, oranges, whole-wheat products, liver, asparagus, beets, broccoli, brussels sprouts, and spinach.
  Folic acid helps your body produce and maintain new cells, and also helps prevent changes to DNA that may lead to cancer.

SUMMARY:
For many years there is a lack of large randomized controlled trials that study the effect of low dose prednisone in women with RPL and thus the evidence of a probable efficacy of prednisone in RPL women remains limited and unclear. As the ESHRE recommended in 2018 (2) we aim to assess the effect of such treatment in a large trial that includes unexplained and abnormal autoimmune profile RPL patients. we also aim to assess the side effects of the treatment in RPL pregnant women.

DETAILED DESCRIPTION:
Recurrent pregnancy loss (RPL) was defined recently by the European society of human reproduction and embryology (ESHRE) as the loss of two or more pregnancies that occur after spontaneous conception and assisted reproductive technology excluding ectopic, molar pregnancies and implantation failure (1,2). The exact prevalence of RPL is difficult to estimate but most studies including the American society for reproductive medicine (ASRM) repost that RPL affects 5% of women. In approximately half of the women with RPL the etiology will remain unexplained while in the remaining half the cause will be defined as one or more of the following, genetic factors, anatomic factors, endocrine factors, autoimmune and infectious (1,3-6). 15% of patients with RPL are diagnosed with antiphospholipid syndrome which is considered as an autoimmune disease (7,8). The ESHRE and ASRM guidelines recommend treatment of prophylactic doses of unfractionated heparin and low-dose aspirin for RPL women with high titers of antiphospholipid antibodies. For RPL women with the remaining immunological conditions glucocorticosteroids, IvIg , TNF inhibitors, and G-CSF treatment are not evidence-based but can be given in research context (1,4,8). Glucocorticosteroids are drugs that reduce inflammation by blocking the expression of proinflammatory cytokines. They suppress the activity of T cells and decrease cytokines levels- IL6, IL1β, TNFα. This drug is a known treatment for inflammatory diseases including asthma, Crohn's disease, and rheumatoid arthritis (9,10). In a recent review in 2017 Bandoli et al (11) summarized that corticosteroids are often necessary to control the symptoms of various medical conditions in pregnancy, including rheumatoid arthritis, systemic lupus erythematosus, and inflammatory bowel disease. Investigations into adverse pregnancy and birth outcomes following corticosteroid exposure have lacked adequate exploration into confounding by disease or disease severity. The evidence for cleft palate alone is not sufficient to summarize. The estimated risk of cleft lip with or without cleft palate from corticosteroid exposure has weakened over time, and no study published after 2003 has reported a statistically significant risk estimate. This review does not find sufficient evidence to support an increased risk of preterm birth, low birth weight, or preeclampsia following systemic corticosteroid use in pregnancy. There is insufficient evidence to determine whether systemic corticosteroids are linked to gestational diabetes mellitus.

Recently, a few studies were conducted with different protocols to investigate the impact of steroid therapy on women with RPL. Eight studies had reported a positive effect of prednisone on live birth rate. Hasegawa et al (12) found a significantly effective live birth rate of 76.5% compared to 8.3% (p<0.01) in 17 treated RPL patients with antiphospholipid antibody with Prednisolone (40 mg/day) as soon as pregnancy was diagnosed, for at least 4 weeks together with low dose Aspirin (81 mg/day) until delivery, and 12 untreated patients respectively. They also found decreased antiphospholipid antibody titer and lower IUGR rate in the study group (30.8% compared to 83.3%, p<0.05). Reznikoff et al (13) reported on the influence of steroid therapy combined with low dose Aspirin on the live birth rate in RPL autoantibody negative pregnant women. In his study he found a 90.7% live birth rate among 214 women treated with Prednisone (20 mg/day) in the first trimester only and low dose Aspirin (100 mg/day) for 7 months, compared with 74.6% birth rate among 63 women receiving aspirin alone (p<0.001). Bansal et al (14) claimed in his review that a combination of Prednisone with low-dose aspirin can be efficient in preventing RPL, mainly in the first trimester of pregnancy, especially in women with non-APAS autoimmunity. Ogasawara et al (15) reported about a birth of a healthy baby to a woman who experienced 10 unexplained first trimester miscarriages after receiving intra-uterine Prednisolone (8 mg of 2 ml of solumedrol) 2-3 days before ovulation and aspirin (40 mg/day) from 4 until 36 weeks of gestation. Gomaa et al (16) reported an ongoing pregnancy beyond 20 weeks of gestation in 70.3 % of women in the prednisolone treatment group and only 9.2% in the placebo group. In three different studies, Quenby et al have shown a positive effect of steroid therapy on reducing the number of uterine NK cells (from 14% before treatment to 9% after, p=0.0004) by given Prednisone (20 mg/day, from day 1 to 21 of the menstrual cycle) to 28 women with RPL and high number of uterine NK cells(17). She reported about a birth of a healthy baby to a woman that suffered from 19 consecutive miscarriages after receiving prednisolone (20 mg/day) for 6 months prior to conception until 5 weeks gestation(18). In a latest study, a 60% and 40% live birth rate was reported in a small treatment and placebo group respectively both with no pregnancy complications nor serious adverse fetal outcomes, although the results weren't statistically significant (19).

Three studies have shown a probable positive effect of prednisone on birth life rate but have reported complications. Tempefar et al (20)reported 77% and 35% live birth rates in a 52 RPL women group who received a combination of Prednisone (20 mg/day), Progesterone (20 mg/day) for the first 12 weeks, Aspirin (100 mg/day) until 38 weeks of gestation and Folic-acid (5 mg) every second day throughout the pregnancy, and in a 52 RPL women control group respectively. Complications including nausea, depression, and tachycardia were observed. Cushing's disease and IUGR were not observed, neither a difference of mean birth weight nor preterm birth rate. Kumar et al (21)suggested that steroid therapy restricted to the preconception and early pregnancy for women with non-APAS autoimmunity may improve the outcome of the pregnancy. However, Kumar noted that steroid therapy during pregnancy is associated with a higher risk for preterm labor secondary to rupture of membranes and to the development of preeclampsia and gestational diabetes. Wang et al (22) who used high doses Prednisone (40-50 mg/day), reported on the increased risk of preterm labor and recommended not to used high doses prednisone for RPL women.

Two studies didn't show improvement of steroid therapy in the outcome of pregnancy. Laskin et al (23) published a study on 773 women with RPL and autoantibodies (antinuclear, anti-DNA, antilymphocyte, anticardiolipin and lupus anticoagulant antibodies). The women were divided into treatment group (received high dose Prednisone 0.5-0.8 mg/kg/day + Aspirin 100 mg/day) and to a placebo group. No significant difference in live birth was reported between the two groups. However, preterm labor (62% and 12%, p<0.01), hypertension (13%&5%, p=0.05) and gestational diabetes (15%&5%, p=0.02) were more common in the treatment group. Empson et al (24) reviewed the influence of prednisone and aspirin treatment for RPL women with antiphospholipid antibody or lupus anticoagulant. He reported higher rates of prematurity and gestational diabetes in the steroid treatment group without an improvement in pregnancy outcome.

To summarise for many years there is a lack of large randomized controlled trials that study the effect of low dose prednisone in women with RPL and thus the evidence of a probable efficacy of prednisone in RPL women remains limited and unclear. As the ESHRE recommended in 2018 (2) we aim to assess the effect of such treatment in a large trial that includes unexplained and abnormal autoimmune profile RPL patients. we also aim to assess the side effects of the treatment in RPL pregnant women.

ELIGIBILITY:
Inclusion Criteria:

* Patients with unexplained RPL.
* Patients with abnormal immunological profile, including ANA, RF, anti-DNA, antilymphocyte, anticardiolipin, antithyroid and lupus anticoagulant antibodies that have no other clinical manifestation.
* Women with three or more pregnancy losses (before 24 weeks of gestation) who referred to the RPL clinic in Soroka hospital.
* An age above 25 years.
* The women agreed to participate in the study and signed on a consent form.
* women with index pregnancy.

Exclusion Criteria:

* Presence of any genetic impairment, Mullerian anomaly, endocrine or metabolic disorders, or a luteal-phase defect (as determined by a timed endometrial biopsy).
* Diabetes mellitus diagnosed by symptoms of diabetes plus random glucose concentration≥ 200mg/dL or fasting plasma glucose≥ 126mg/dL or hemoglobin A1C≥5.8% or 2-h plasma glucose≥ 200mg/dL during an oral glucose tolerance test.
* Previously untreated tuberculosis, as determined by an abnormal chest film in the previous year or a positive tuberculin skin test.
* Prednisone therapy during pregnancy for other reasons.
* Sensitivity to prednisone.

Ages: 25 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 242 (Estimated)
Dates: Start 2020-12 (Estimated); Primary Completion 2021-07 (Estimated); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
Live birth | through study completion, an average of 1 year.
  birth that occurs after 24 weeks of gestation.
Pregnancy loss | through study completion, an average of 1 year.
  birth that occurs up to 24 weeks of gestation.

CONTACTS AND LOCATIONS:
Locations (1):
- Soroka Medical Center, Beersheba, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] ESHRE Guideline Group on RPL; Bender Atik R, Christiansen OB, Elson J, Kolte AM, Lewis S, Middeldorp S, Nelen W, Peramo B, Quenby S, Vermeulen N, Goddijn M. ESHRE guideline: recurrent pregnancy loss. Hum Reprod Open. 2018 Apr 6;2018(2):hoy004. doi: 10.1093/hropen/hoy004. eCollection 2018. PMID 31486805
- [Background] (2) Mehta S, Gupta B. Recurrent Pregnancy Loss. 2018 Apr 20,.
- [Background] Ford HB, Schust DJ. Recurrent pregnancy loss: etiology, diagnosis, and therapy. Rev Obstet Gynecol. 2009 Spring;2(2):76-83. PMID 19609401
- [Background] Practice Committee of the American Society for Reproductive Medicine. Evaluation and treatment of recurrent pregnancy loss: a committee opinion. Fertil Steril. 2012 Nov;98(5):1103-11. doi: 10.1016/j.fertnstert.2012.06.048. Epub 2012 Jul 24. PMID 22835448
- [Background] Gabbai D, Harlev A, Friger M, Steiner N, Sergienko R, Kreinin A, Bashiri A. Pregnancy outcomes among patients with recurrent pregnancy loss and uterine anatomic abnormalities. J Perinat Med. 2018 Sep 25;46(7):728-734. doi: 10.1515/jpm-2016-0411. No abstract available. PMID 28742523
- [Background] Kabessa M, Harlev A, Friger M, Sergienko R, Litwak B, Koifman A, Steiner N, Bashiri A. Pregnancy outcomes among patients with recurrent pregnancy loss and chromosomal aberration (CA) without PGD. J Perinat Med. 2018 Sep 25;46(7):764-770. doi: 10.1515/jpm-2016-0408. No abstract available. PMID 28672755
- [Background] El Hachem H, Crepaux V, May-Panloup P, Descamps P, Legendre G, Bouet PE. Recurrent pregnancy loss: current perspectives. Int J Womens Health. 2017 May 17;9:331-345. doi: 10.2147/IJWH.S100817. eCollection 2017. PMID 28553146
- [Background] Bashiri A, Gete S, Mazor M, Gete M. [Recurrent pregnancy loss--evaluation and treatment]. Harefuah. 2011 Nov;150(11):852-6, 875. Hebrew. PMID 22428207
- [Background] Barnes PJ. How corticosteroids control inflammation: Quintiles Prize Lecture 2005. Br J Pharmacol. 2006 Jun;148(3):245-54. doi: 10.1038/sj.bjp.0706736. PMID 16604091
- [Background] Feldman PA, Wolfson D, Barkin JS. Medical management of Crohn's disease. Clin Colon Rectal Surg. 2007 Nov;20(4):269-81. doi: 10.1055/s-2007-991026. PMID 20011423
- [Background] Bandoli G, Palmsten K, Forbess Smith CJ, Chambers CD. A Review of Systemic Corticosteroid Use in Pregnancy and the Risk of Select Pregnancy and Birth Outcomes. Rheum Dis Clin North Am. 2017 Aug;43(3):489-502. doi: 10.1016/j.rdc.2017.04.013. PMID 28711148
- [Background] Hasegawa I, Takakuwa K, Goto S, Yamada K, Sekizuka N, Kanazawa K, Tanaka K. Effectiveness of prednisolone/aspirin therapy for recurrent aborters with antiphospholipid antibody. Hum Reprod. 1992 Feb;7(2):203-7. doi: 10.1093/oxfordjournals.humrep.a137617. PMID 1577931
- [Background] Reznikoff-Etievant MF, Cayol V, Zou GM, Abuaf N, Robert A, Johanet C, Milliez J. Habitual abortions in 678 healthy patients: investigation and prevention. Hum Reprod. 1999 Aug;14(8):2106-9. doi: 10.1093/humrep/14.8.2106. PMID 10438434
- [Background] Bansal AS, Bajardeen B, Thum MY. The basis and value of currently used immunomodulatory therapies in recurrent miscarriage. J Reprod Immunol. 2012 Jan;93(1):41-51. doi: 10.1016/j.jri.2011.10.002. Epub 2011 Dec 21. PMID 22196105
- [Background] Ogasawara M, Aoki K. Successful uterine steroid therapy in a case with a history of ten miscarriages. Am J Reprod Immunol. 2000 Oct;44(4):253-5. doi: 10.1111/j.8755-8920.2000.440411.x. PMID 11076099
- [Background] Gomaa MF, Elkholy AG, El-Said MM, Abdel-Salam NE. Combined oral prednisolone and heparin versus heparin: the effect on peripheral NK cells and clinical outcome in patients with unexplained recurrent miscarriage. A double-blind placebo randomized controlled trial. Arch Gynecol Obstet. 2014 Oct;290(4):757-62. doi: 10.1007/s00404-014-3262-0. Epub 2014 May 13. PMID 24818590
- [Background] Quenby S, Kalumbi C, Bates M, Farquharson R, Vince G. Prednisolone reduces preconceptual endometrial natural killer cells in women with recurrent miscarriage. Fertil Steril. 2005 Oct;84(4):980-4. doi: 10.1016/j.fertnstert.2005.05.012. PMID 16213853
- [Background] Quenby S, Farquharson R, Young M, Vince G. Successful pregnancy outcome following 19 consecutive miscarriages: case report. Hum Reprod. 2003 Dec;18(12):2562-4. doi: 10.1093/humrep/deg502. PMID 14645171
- [Background] Tang AW, Alfirevic Z, Turner MA, Drury JA, Small R, Quenby S. A feasibility trial of screening women with idiopathic recurrent miscarriage for high uterine natural killer cell density and randomizing to prednisolone or placebo when pregnant. Hum Reprod. 2013 Jul;28(7):1743-52. doi: 10.1093/humrep/det117. Epub 2013 Apr 12. PMID 23585559
- [Background] Tempfer CB, Kurz C, Bentz EK, Unfried G, Walch K, Czizek U, Huber JC. A combination treatment of prednisone, aspirin, folate, and progesterone in women with idiopathic recurrent miscarriage: a matched-pair study. Fertil Steril. 2006 Jul;86(1):145-8. doi: 10.1016/j.fertnstert.2005.12.035. Epub 2006 May 23. PMID 16716321
- [Background] Kumar A. Immunomodulation in recurrent miscarriage. J Obstet Gynaecol India. 2014 Jun;64(3):165-8. doi: 10.1007/s13224-014-0541-4. Epub 2014 May 8. PMID 24966498
- [Background] Wang SW, Zhong SY, Lou LJ, Hu ZF, Sun HY, Zhu HY. The effect of intravenous immunoglobulin passive immunotherapy on unexplained recurrent spontaneous abortion: a meta-analysis. Reprod Biomed Online. 2016 Dec;33(6):720-736. doi: 10.1016/j.rbmo.2016.08.025. Epub 2016 Sep 16. PMID 27720163
- [Background] Laskin CA, Bombardier C, Hannah ME, Mandel FP, Ritchie JW, Farewell V, Farine D, Spitzer K, Fielding L, Soloninka CA, Yeung M. Prednisone and aspirin in women with autoantibodies and unexplained recurrent fetal loss. N Engl J Med. 1997 Jul 17;337(3):148-53. doi: 10.1056/NEJM199707173370302. PMID 9219700
- [Background] Empson M, Lassere M, Craig J, Scott J. Prevention of recurrent miscarriage for women with antiphospholipid antibody or lupus anticoagulant. Cochrane Database Syst Rev. 2005 Apr 18;2005(2):CD002859. doi: 10.1002/14651858.CD002859.pub2. PMID 15846641